CLINICAL TRIAL: NCT02204527
Title: Supplementation of Vitamin D in Patients With Type 2 Diabetes and Hypertension: Randomized Clinical Trial
Brief Title: Supplementation of Vitamin D in Patients With Type 2 Diabetes and Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Mirela Jobim de Azevedo, Mirela Jobim Azevedo, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 140415
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension
Keywords: hypertension; diabetes mellitus; vitamin D
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This study was a randomized, double-blind, placebo-controlled clinical trial on 40 outpatients with hypertension and type 2 diabetes were recruited.
  Patients were allocated into two equal groups of 20 by computer-generated randomly permutated codes. the subjects were randomly assigned to 1 of 2 groups: Group 1 received a single dose (100.000 IU) of oral supplementation with cholecalciferol (vitamin D3). Group 2 received matching placebo capsules containing microcrystalline cellulose.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D3 (Experimental): supplementation of 100.000 IU of vitamin D3
  Interventions: Dietary Supplement: supplementation of 100.000 IU of vitamin D3
- Placebo pill (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: placebo pill

INTERVENTIONS:
Dietary Supplement: supplementation of 100.000 IU of vitamin D3 — supplementation of vitamin D ( with 2 pills of Addera D3 (50.000IU each pill))
  Other Names: supplementation of 100.000 IU of vitamin D3: Addera D3 (50.000IU each pill)
  Arms: vitamin D3
Dietary Supplement: placebo pill — Placebo
  Other Names: Placebo
  Arms: Placebo pill

SUMMARY:
In patients with type 2 diabetes, the effects on blood pressure of vitamin D has been shown to be variable. Thus, the goal of this proposal is to evaluate the effect of vitamin D supplementation in patients with type 2 diabetes and hypertension

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* hypovitaminosis D
* hypertension

Exclusion Criteria:

* pregnant or lactating
* patients using vitamin D supplementation
* using drugs that interfere on vitamin D metabolism (corticosteroids, anticonvulsants)
* illicit drug use
* diseases such as chronic renal failure (serum creatinine greater than 2.0 mg/dl)
* liver cirrhosis
* alcoholism
* dementia
* malignant disease that compromises the 5-year survival,
* digestive tract (malabsorption) diseases
* BMI> 40 kg / m2

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Ambulatory Blood pressure monitoring | up to 24 hours
  Blood pressure will be assessed by Ambulatory Blood Pressure Monitoring before and after vitamin D supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- HCPA, Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] de Paula TP, Moreira JSR, Sperb LF, Muller MEP, Steemburgo T, Viana LV. Efficacy of single-dose cholecalciferol in the blood pressure of patients with type 2 diabetes, hypertension and hypovitaminoses D. Sci Rep. 2020 Nov 12;10(1):19611. doi: 10.1038/s41598-020-76646-6. PMID 33184328